CLINICAL TRIAL: NCT00926939
Title: Technological Innovations in Behavioral Treatments for Cigarette Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jesse Dallery, Principal Investigator, National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA023469 (NIH); R01DA023469 (NIH)
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Cigarette Smoking
Keywords: Cigarette; Nicotine; Smoking; Contingency Management; Voucher reinforcement; Smoking Abstinence; Internet-based treatment
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abstinence Contingent (AC) (Experimental): This group will receive vouchers contingent on smoking reduction and smoking abstinence (confirmed through video submissions). Abstinence is defined as a CO sample of 4ppm or less.
  Interventions: Behavioral: Reinforcement for the abstinence of smoking
- Submission Contingent (SC) (Experimental): This group receives vouchers for submitting videos of their CO breath test.
  Interventions: Behavioral: Reinforcement for submission of videos with CO sample

INTERVENTIONS:
Behavioral: Reinforcement for the abstinence of smoking — Participants in this intervention group will receive vouchers contingent upon a CO sample of 4ppm or less.
  Arms: Abstinence Contingent (AC)
Behavioral: Reinforcement for submission of videos with CO sample — This intervention group will receive vouchers contingent on their submission of videos of their CO breath tests.
  Arms: Submission Contingent (SC)

SUMMARY:
The purpose of the study is to evaluate a sustainable and broadly accessible treatment delivery model (Motiv8) for smoking cessation based on abstinence-reinforcement.

DETAILED DESCRIPTION:
Smokers are randomly assigned to one of two groups: an Abstinence Contingent (AC) group and a Submission Contingent (SC) group. The AC group receives vouchers for abstaining from smoking (measured by a carbon monoxide monitor and confirmed through video-submission), and the SC group receives vouchers for submitting videos of their carbon monoxide breath tests. Both groups take videos of their CO-monitoring on a secure website designed for the study, as well as receive standard care counseling and education related to smoking cessation. The main intervention lasts four weeks, and a three-week maintenance phase will follow. Assessments will be conducted at intake, week four (end of the main treatment phase), and at three and six months after the intervention period is completed

ELIGIBILITY:
Inclusion Criteria:

* Self-reported smoker
* Permission to contact applicant by phone
* Ability to use the internet

Exclusion Criteria:

* Self-report of a history of or current severe or unstable medical or psychiatric illness that would interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
CO sample of ≤ 4ppm | 4 weeks, 7 weeks during intervention; 3 months and 6 months after intervention
Participant reporting not smoking, not even a puff in the last 7 days. | 4 weeks, 7 weeks during intervention; 3 months and 6 months after intervention

SECONDARY OUTCOMES:
Twice-daily breath CO samples obtained during treatment period. | First 4 weeks of treatment
The longest duration of sustained abstinence based on the twice-daily breath samples during the treatment period. | First 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dallery, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- National Development and Research Institutes, New York, New York, United States

REFERENCES:
- See also: Study website — http://www.psych.ufl.edu/~ufsmokelab